CLINICAL TRIAL: NCT01558297
Title: Internet Treatment for Weight Loss in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rachel D. Barnes, Associate Research Scienist, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1106008713; 1K23DK092279-01 (NIH)
Record Dates: First submitted 2012-03-15; First posted 2012-03-20 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity | interventions — Motivational Interviewing; Nutrition Assessment; Therapeutics; Physicians, Primary Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing
- Nutritional Counseling (Active Comparator)
  Interventions: Behavioral: Nutritional Counseling
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual with primary care physician

INTERVENTIONS:
Behavioral: Motivational Interviewing — 5 sessions of motivational interviewing over a period of 3 months.
  Arms: Motivational Interviewing
Behavioral: Nutritional Counseling — 5 sessions of nutritional counseling over a period of 3 months.
  Arms: Nutritional Counseling
Behavioral: Treatment as usual with primary care physician — Participants will be encouraged to continue their care with their primary care physician.
  Arms: Treatment as usual

SUMMARY:
This study will test the effectiveness of two distinct treatments for weight loss:

1. Motivational Interviewing
2. Nutritional Counseling. These treatments will be compared to Treatment as Usual. Participants will be recruited through local primary care offices.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-55
* Daily access to internet and phone

Exclusion Criteria:

* Co-existing physical and/or psychiatric conditions that require more significant treatment (e.g., bipolar disorder, psychotic illnesses), and/or require more intensive treatment or hospitalization (e.g., suicidality, severe mood disorders)
* Meets criteria for current substance abuse or dependence
* Currently receiving psychiatric, psychological, behavioral, or pharmacologic treatment that is known to affect weight or eating
* Pregnant, breastfeeding, or plans to become pregnant during the treatment period
* Cardiac disease, including ischemic heart disease, congestive heart failure, conduction abnormalities, or a history of heart attack
* Serious neurologic illnesses (e.g., seizure history) or medical illnesses (e.g., impaired hepatic or renal function)
* Uncontrolled diabetes, thyroid conditions, or hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Barnes, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Result] Barnes RD, White MA, Martino S, Grilo CM. A randomized controlled trial comparing scalable weight loss treatments in primary care. Obesity (Silver Spring). 2014 Dec;22(12):2508-16. doi: 10.1002/oby.20889. Epub 2014 Oct 9. PMID 25298016
- [Derived] Wiedemann AA, Baumgardt SS, Ivezaj V, Kerrigan SG, Lydecker JA, Grilo CM, Barnes RD. Getting a head start: identifying pretreatment correlates associated with early weight loss for individuals participating in weight loss treatment. Transl Behav Med. 2021 Feb 11;11(1):236-243. doi: 10.1093/tbm/ibz149. PMID 31816053

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interviewing | Nutritional Counseling | Treatment as Usual
Started | 30 | 29 | 30
Completed | 28 | 27 | 29
Not Completed | 2 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Chi-square for categorical variables and ANOVAs for continuous variables.
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing | Nutritional Counseling | Treatment as Usual | Total
Number analyzed (Participants) | 30 | 29 | 30 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.07 (9.97) | 48.93 (11.59) | 47.77 (10.05) | 47.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 24 | 68
  Male | 6 | 9 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 3 | 7 | 18
  White | 19 | 22 | 21 | 62
  More than one race | 3 | 4 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Body Weight in Pounds.
Description: Body weight lost in pounds measured 1.5 months after first treatment session.
Time Frame: 1.5 months after treatment start (Baseline)
Population: Intent-to-treat data are presented, with the last observation carried forward, and outliers beyond 3 standard deviations replaced with highest recorded value within the 3 standard deviation range.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Motivational Interviewing | Nutritional Counseling | Treatment as Usual
Number analyzed (Participants) | 30 | 29 | 30
pounds | -3.1 (4.6) | -3.4 (5.2) | 0.1 (3.5)

2. Primary Outcome: Body Weight in Pounds.
Description: Body weight lost in pounds measured 3 months after first treatment session.
Time Frame: 3 months after treatment start (Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Motivational Interviewing | Nutritional Counseling | Treatment as Usual
Number analyzed (Participants) | 30 | 29 | 30
pounds | -3.3 (6.5) | -4.9 (6.1) | -0.4 (6.2)

3. Primary Outcome: Body Weight in Pounds.
Description: Body weight lost in pounds measured 6 months after first treatment session (3 month follow-up after active treatment ends).
Time Frame: 6 months after treatment start (Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Motivational Interviewing | Nutritional Counseling | Treatment as Usual
Number analyzed (Participants) | 30 | 29 | 30
pounds | -2.6 (8.7) | -5.7 (9.0) | 0.4 (7.2)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Motivational Interviewing | Nutritional Counseling | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Treatment as Usual (TAU) was subsequently referred to as Usual Care (UC) when the study results were disseminated because the literature evolved regarding treatment terms. UC more accurately reflect the condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No